CLINICAL TRIAL: NCT00005968
Title: A Multicenter Phase II Trial of MGI-114 in Patients With Stage IV Malignant Melanoma
Brief Title: Irofulven in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 99-0468.cc; UCHSC-99468; NCI-T99-0070
Record Dates: First submitted 2000-07-05; First posted 2004-06-21 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2002-12

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — irofulven

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and duration of response in patients with stage IV malignant melanoma treated with 6-hydroxymethylacylfulvene. II. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive 6-hydroxymethylacylfulvene IV over 5 minutes on days 1-5. Treatment repeats every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after completion of course 2 receive additional courses. Patients are followed every 3 months for 5 years, and then annually thereafter until death.

PROJECTED ACCRUAL: Approximately 16-35 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IV malignant melanoma No prior chemotherapy OR No more than 1 prior chemotherapy containing regimen Measurable disease Brain metastasis allowed if adequately treated

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Hemoglobin at least 10 g/dL WBC at least 4,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) ALT/AST no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: See Disease Characteristics Recovered from any prior therapy No other concurrent therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rene Gonzalez, MD, Study Chair — University of Colorado, Denver
Locations (5):
- United States (5):
  - John Wayne Cancer Institute, Santa Monica, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Lutheran General Hospital, Park Ridge, Illinois
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri